CLINICAL TRIAL: NCT06404411
Title: A Study of the Efficacy of Aerobic Exercise Based on Cardiopulmonary Exercise Test in the Rehabilitation of Patients With COVID-19-Related Myocardial Injury
Brief Title: The Efficacy of Aerobic Exercise in the Rehabilitation of Patients With COVID-19-Related Myocardial Injury
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chengdu Sport University (Other)
Responsible Party: Principal Investigator, Ping Yang, Clinical Professor, Chengdu Sport University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024058H
Record Dates: First submitted 2024-05-07; First posted 2024-05-08 (Actual); Last update posted 2024-05-13 (Actual); Status verified 2024-05

CONDITIONS: Long COVID; Myocardial Injury
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention group (Experimental)
  Interventions: Other: Assigned interventions; Other: conventional rehabilitation
- control group (Active Comparator)
  Interventions: Other: conventional rehabilitation

INTERVENTIONS:
Other: Assigned interventions — Combined aerobic endurance exercise in the control group: individualized exercise prescription, including 5-10 minutes of pre-exercise dynamic stretching and warm-up, 10-30 minutes of formal aerobic exercise, and 5-10 minutes of post-exercise stretching, formal aerobic exercise using a power bike starting from low-intensity and gradually increasing to medium-high-intensity, with a frequency of five times per week.
  Other Names: aerobic endurance exercise
  Arms: intervention group
Other: conventional rehabilitation — Adoption of conventional rehabilitation, drug therapy, enhanced nutritional support and other conventional treatment

SUMMARY:
A study of the efficacy of aerobic exercise based on cardiopulmonary exercise test in the rehabilitation of patients with COVID-19-related myocardial injury

ELIGIBILITY:
Inclusion Criteria:

1. Between the ages of 18 and 65 years;
2. A history of new coronavirus infection;
3. Patients with a clinical diagnosis of COVID-19-related myocardial injury;
4. In the late stages of recovery from COVID-19-related myocardial injury, at least 3 months after diagnosis;
5. Negative cardiopulmonary exercise test;
6. After completing respiratory rehabilitation at our hospital in the previous period;
7. Normal blood biomarker tests and essentially normal 2D-STE, normal left ventricular systolic function, no spontaneous or inducible arrhythmias on electrocardiographic monitoring, and the patient's clinical status is stable, with most of the symptoms in significant remission, and the daily still activities are intolerant or do not reach the pre-disease exercise level;
8. Classification of nyha heart function of class I or II;
9. Voluntarily sign the informed consent form;
10. Not participating in other clinical trials.

Exclusion Criteria:

1. a previous history of coronary atherosclerotic heart disease and heart failure;
2. a combination of severe arrhythmia or cardiogenic shock;
3. a combination of severe hypertension, hypertrophic cardiomyopathy, valvular disease of moderate or greater severity, acute myocarditis or pericarditis;
4. a combination of any disease that severely affects limb movement, such as musculoskeletal disorders or severe hepatic or renal insufficiency
5. a combination of progressive malignant tumors, infectious diseases, bleeding disorders, autoimmune diseases, etc;
6. those who have serious mental illness and are unable to cooperate
7. those with incomplete clinical data;
8. those who have dropped out or terminated the trial by themselves.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-06-30 (Estimated); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
VO2peak | 12 weeks
  All subjects were exercised in a plank fashion, using a modified Bruce protocol, in which the speed and incline were gradually increased by one level every 3 minutes during the test until the end of the exercise to reach the subject's sub-extreme volume of exercise, so that peak metabolic equivalents (METpeak), peak oxygen uptake (peak oxygen uptake, VO2peak), anaerobic threshold ( anaerobic threshold, AT), peak minute ventilation (VEpeak), breath reserve (BR), and peak oxygen pulse (VO2/HRpeak).

SECONDARY OUTCOMES:
METpeak | 12 weeks
  All subjects were exercised in a plank fashion, using a modified Bruce protocol, in which the speed and incline were gradually increased by one level every 3 minutes during the test until the end of the exercise to reach the subject's sub-extreme volume of exercise, so that peak metabolic equivalents (METpeak), peak oxygen uptake (peak oxygen uptake, VO2peak), anaerobic threshold ( anaerobic threshold, AT), peak minute ventilation (VEpeak), breath reserve (BR), and peak oxygen pulse (VO2/HRpeak).
AT | 12 weeks
  All subjects were exercised in a plank fashion, using a modified Bruce protocol, in which the speed and incline were gradually increased by one level every 3 minutes during the test until the end of the exercise to reach the subject's sub-extreme volume of exercise, so that peak metabolic equivalents (METpeak), peak oxygen uptake (peak oxygen uptake, VO2peak), anaerobic threshold ( anaerobic threshold, AT), peak minute ventilation (VEpeak), breath reserve (BR), and peak oxygen pulse (VO2/HRpeak).
VEpeak | 12 weeks
  All subjects were exercised in a plank fashion, using a modified Bruce protocol, in which the speed and incline were gradually increased by one level every 3 minutes during the test until the end of the exercise to reach the subject's sub-extreme volume of exercise, so that peak metabolic equivalents (METpeak), peak oxygen uptake (peak oxygen uptake, VO2peak), anaerobic threshold ( anaerobic threshold, AT), peak minute ventilation (VEpeak), breath reserve (BR), and peak oxygen pulse (VO2/HRpeak).
BR | 12 weeks
  All subjects were exercised in a plank fashion, using a modified Bruce protocol, in which the speed and incline were gradually increased by one level every 3 minutes during the test until the end of the exercise to reach the subject's sub-extreme volume of exercise, so that peak metabolic equivalents (METpeak), peak oxygen uptake (peak oxygen uptake, VO2peak), anaerobic threshold ( anaerobic threshold, AT), peak minute ventilation (VEpeak), breath reserve (BR), and peak oxygen pulse (VO2/HRpeak).
VO2/HRpeak | 12 weeks
  All subjects were exercised in a plank fashion, using a modified Bruce protocol, in which the speed and incline were gradually increased by one level every 3 minutes during the test until the end of the exercise to reach the subject's sub-extreme volume of exercise, so that peak metabolic equivalents (METpeak), peak oxygen uptake (peak oxygen uptake, VO2peak), anaerobic threshold ( anaerobic threshold, AT), peak minute ventilation (VEpeak), breath reserve (BR), and peak oxygen pulse (VO2/HRpeak).
Six-minute walk test distance, 6MWD | 12 weeks
  Select a 30-meter-long section of the corridor and post the location of the starting and ending points. Subjects were instructed to walk back and forth through the 30-meter passageway for 6 minutes, covering the longest distance as fast as they could.
SDNN | 12 weeks
  Data were captured for each subject at baseline, after 12 weeks of exercise intervention, using an ambulatory electrocardiogram for 24 hours continuously. Each phase was worn once, for a continuous 24-hour period.
SDANN | 12 weeks
  Data were captured for each subject at baseline, after 12 weeks of exercise intervention, using an ambulatory electrocardiogram for 24 hours continuously. Each phase was worn once, for a continuous 24-hour period.
RMSSD | 12 weeks
  Data were captured for each subject at baseline, after 12 weeks of exercise intervention, using an ambulatory electrocardiogram for 24 hours continuously. Each phase was worn once, for a continuous 24-hour period.
physical composite scale，PCS | 12 weeks
  The SF-12v2 is a shortened version of the scale developed based on the SF-36, which is comprehensive, simple, and less time-consuming, and is used to evaluate subjects' quality of life with 12 entries and 8 dimensions: general health, somatic functioning, somatic functioning, bodily pain, vitality, social functioning, affective functioning, and mental health. The higher the score, the better the quality of life and functional status of the patient.
mental health composite scale，MCS | 12 weeks
  The SF-12v2 is a shortened version of the scale developed based on the SF-36, which is comprehensive, simple, and less time-consuming, and is used to evaluate subjects' quality of life with 12 entries and 8 dimensions: general health, somatic functioning, somatic functioning, bodily pain, vitality, social functioning, affective functioning, and mental health. The higher the score, the better the quality of life and functional status of the patient.